CLINICAL TRIAL: NCT00491361
Title: Psychometric Study of the Chinese Versions of the Swanson, Nolan, and Pelham, Version IV (SNAP-IV) Scale and Strengths Difficulties Questionnaire.
Brief Title: Chinese Versions of the Swanson, Nolan, and Pelham, Version IV (SNAP-IV) Scale and Strengths Difficulties Questionnaire.
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 9461700519; NTUH95-301 (Other: National Taiwan University Hospital)
Record Dates: First submitted 2007-06-23; First posted 2007-06-26 (Estimated); Last update posted 2012-11-14 (Estimated); Status verified 2008-08

CONDITIONS: Attention-deficit/Hyperactivity Disorder
Keywords: ADHD, SNAP-IV, SDQ, ASRS, reliability, validity
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

SUMMARY:
Background: Attention-Deficit/Hyperactivity Disorder (ADHD) is a common childhood-onset neuropsychiatric disorder (7.5% in Taiwan) with great impact on individual, family, and society. The diagnosis of ADHD is mainly based on clinical interview of parents and children with assistance of teachers' reports. Self-administered rating scales are useful for screening, assistance of diagnosis, and measurement of symptom changes over time or due to treatment effect. The goals of this study are to establish the norms and psychometric properties of the Chinese version of teacher and parent forms of the Swanson, Nolan, and Pelham, version IV (SNAP-IV) and the teacher, parent, and student forms of the Strengths and Difficulties Questionnaire (SDQ) for future studies on ADHD in Taiwanese populations.

Subjects and Methods: This is a cross-sectional, school-based survey with a multi-stage sampling method. The participants include a school-based sample of 3534 first to eighth graders was recruited from four areas: Taipei City, Taoyuan County, Tainan City and Chiayi County. Among them, 200students will be reassessed at 2-week interval for the test-retest reliability study. The instruments comprise the Chinese version of Child Behavioral Checklist (CBCL), SDQ, SNAP-IV, and Adult ADHD Rating Scale. The informants include student participants older than 10 years old, their parents, and teachers. The main statistical methods include Pearson correlation, intraclass correlation, Chronbach's α for internal consistency, and mixed model to address lack of independence within the same classes and schools.

Anticipated Goals: We expect that this study will reach the following objectives:

1. to obtain the primitive information about the prevalence of ADHD symptoms and emotional/behavioral problems among children and adolescents in Taipei and Yun-Ling;
2. to enhance the awareness of school teachers and counselors about ADHD and other behavioral/emotional problems among students;
3. to establish psychometric properties of the Chinese versions of SNAP-IV and SDQ for future use in clinical, school, and research settings.

DETAILED DESCRIPTION:
This protocol was prepared in Chinese

ELIGIBILITY:
Inclusion Criteria:

* School-based subjects: around 3600 grade 1 to grade 8 students aged 6-16 from four sites in Taiwan and their parents (n = 7200)
* Clinical subjects with ADHD: children and adolescents ages 6-16, who are diagnosed with ADHD, IQ >70, parents and teachers consent to completion of questionnaires.

Exclusion Criteria:

* Clinical subjects with ADHD: those who are comorbid with pervasive developmental disorder and/or mental retardation or other severe psychiatric disorders. Oppositional defiant disorder and conduct disorder are not excluded.

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: School-based subjects & Clinical subjects with ADHD
Sampling Method: Non-Probability Sample
Enrollment: 3600 (Actual)
Dates: Start 2005-01; Study Completion 2006-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Shur-Fen Gau, MD, PhD, Principal Investigator — Department of Psychiatry, National Taiwan University Hospital
Locations (1):
- Department of Psychiatry, National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Background] Achenbach, T. M., and Ruffle, T. M. The Child Behavior Checklist and related forms for assessing behavioral/emotional problems and competencies Pediatrics in Review (2000) 21(8):265-71. Becker, A., Woerner, W., Hasselhorn, M., et al. Validation of the parent and teacher SDQ in a clinical sample. European Child & Adolescent Psychiatry (2004) 13 Suppl 2:II11-6. Goodman, R., Ford, T., Corbin, T., et al. Using the Strengths and Difficulties Questionnaire (SDQ) multi-informant algorithm to screen looked-after children for psychiatric disorders. European Child & Adolescent Psychiatry (2004) 13 Suppl 2:II25-31. Yang, H. J., Soong, W. T., Chiang, C. N., et al. Competence and behavioral/emotional problems among Taiwanese adolescents as reported by parents and teachers. Journal of the American Academy of Child & Adolescent Psychiatry (2000) 39(2):232-9.
- [Derived] Gau SS, Lin CH, Hu FC, Shang CY, Swanson JM, Liu YC, Liu SK. Psychometric properties of the Chinese version of the Swanson, Nolan, and Pelham, Version IV Scale-Teacher Form. J Pediatr Psychol. 2009 Sep;34(8):850-61. doi: 10.1093/jpepsy/jsn133. Epub 2008 Dec 12. PMID 19074488